CLINICAL TRIAL: NCT02990416
Title: Phase I/II Trial of the A-dmDT390-bisFv(UCHT1) Fusion Protein in Combination With Ionizing Radiation and Pembrolizumab for the Treatment of Stage IV Melanoma
Brief Title: A-dmDT390-bisFv(UCHT1) Fusion Protein With Ionizing Radiation and Pembrolizumab for the Treatment of Stage IV Melanoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Angimmune LLC (Industry)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDA IND 118558
Record Dates: First submitted 2016-11-28; First posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — A-dmDT390-bisFv(UCHT1) protein; pembrolizumab; Radiation, Ionizing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A-dmDT390-bisFv(UCHT1)/Radiation/Pembrolizumab (Experimental): A-dmDT390-bisFv(UCHT1): 2.5 µg/kg 2x x 4 days, Ionizing Radiation: single treatment on day five of 14-24 Gy to a tumor, Pembrolizumab: 2 mg/kg IV every 3 weeks
  Interventions: Biological: A-dmDT390-bisFv(UCHT1); Biological: Pembrolizumab; Radiation: Ionizing Radiation

INTERVENTIONS:
Biological: A-dmDT390-bisFv(UCHT1) — anti-T cell immunotoxin (antibody targeting CD3 on T-cells tagged with diphtheria toxin without binding domain)
  Other Names: Resimmune® (proposed marketing designation)
Biological: Pembrolizumab — A humanized monoclonal immunoglobulin (Ig) G4 antibody directed against human cell surface receptor PD-1 (programmed death-1 or programmed cell death-1) with potential immune checkpoint inhibitory and antineoplastic activities.
  Other Names: KEYTRUDA
Radiation: Ionizing Radiation — Electromagnetic or corpuscular radiation capable of producing ions, directly or indirectly, in its passage through matter.

SUMMARY:
This study evaluates the effectiveness of adding a single four-day treatment of the fusion protein A-dmDT390-bisFv(UCHT1) - plus single palliative tumor radiation - with standard of care KEYTRUDA (Pembrolizumab) therapy for the treatment of metastatic melanoma. The results will be measured by comparing the combined therapy to historical data of KEYTRUDA alone.

DETAILED DESCRIPTION:
The purpose of this trial is to test the hypothesis that A-dmDT390-bisFv(UCHT1) can act as an immunomodulator of late stage metastatic melanoma when combined with palliative radiation (to induce the priming of activated T cells with tumor antigens) and Pembrolizumab.

A-dmDT390-bisFv(UCHT1), an anti-T cell immunotoxin is currently being studied as a treatment for cutaneous T cell lymphoma and other CD3+ malignant diseases (NCT00611208 and NCT02943642). During the course of this study, data accumulated that A-dmDT390-bisFv(UCHT1) could be acting as an immunomodulator. This was based on the observation that four out of six partial responses converted to complete responses at times ranging between 6 and 24 months following the completion of the 4-day treatment protocol (serum half life ~45 min.) and no other treatment took place. Complete response durations were 4-6+ years.

Checkpoint inhibitors have revolutionized the treatment of certain solid tumors, notably melanoma, NSCLC and renal cancer. Yet the overall response rate remains low and the mechanisms limiting responses have not been elucidated.

Based on the findings that checkpoint inhibitors have higher response rates when the tumor neoantigen burden is higher (over 1 mutation per megabase, Shumacher & Schreiber, 2015) the investigators propose to increase the neoantigen burden by combining two distinct manipulations:

1. Treatment with an anti-CD3 fusion protein Resimmune days 1-4 to induce a 20-fold increase in CD8+ central memory T cells and
2. Treatment with anti-PD1 day 16 and q. 3 weeks to block PD-1/PD-L1 negative regulation on the newly activated T cells (Blake et al., 2015) and to block high levels of PD-1 in the tumor microenvironment (Ahmadzadeh et al., 2009).

Palliative tumor radiation day 5 will provide the tumor antigen release needed to convert the expanded central memory T cells to effector memory T cells.

The study will be a single-arm, uncontrolled phase I/II trial to estimate the safely of the combined treatment and then estimate the efficacy in terms of RECIST 1.1 in patients with stage Stage IV metastatic melanoma. The primary endpoint is the clinical response as defined by progression-free survival (PFS). The second end point will be tolerability to treatment. Secondary end points to be considered are overall survival (OS).

The study is conducted in 2 phases. In phase I (safety), the investigators will enroll 6 patients. In first stage, 25 total patients will be enrolled. Using Simon's two stage minimax design for phase II trials, the investigators plan to enroll a maximum of 63 patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histologically proven stage IV metastatic melanoma consisting of at least two lesions >= 1.5 cm that would not occupy the same radiation field. Patients must be treatment naïve except for treatment with BRAF inhibitors. Patients with melanoma must have an anti-DT titer of <20 μg/ml. Patients with brain metastasis and ocular and mucosal lesions can be enrolled at the discretion of the PI providing that other non-brain and non-ocular metastatic lesions are available as targets for radiation therapy
* Patients must have a performance status of < 2 on Eastern Cooperative Oncology Group scale (see Appendix). Patients must have fully recovered from toxicity of prior therapy with BRAF inhibitors. Adequate bone marrow function will be defined as ANC >750 uL, WBC >1000 uL, platelets >60,000 uL and Hb > 9g/dL
* Patients must have:

  * bilirubin < 1.5 mg/dL,
  * transaminases < 2.5 X ULN,
  * albumin > 3 gm/dL,
  * creatinine < 2.0 mg/dL,
  * adequate pulmonary function by physical exam and pulse oximetry and adequate cardiac reserve (EF > 50% normal).
* Patients must have a normal echocardiogram without any evidence of cardiac chamber hypertrophy, dilatation or hypokinesis. The Sponsor must be provided with copies of these tests before Sponsor will approve enrollment. In addition, the sponsor must receive a list of current medications taken by the patient before Sponsor will approve enrollment.
* Patients must give written informed consent prior to registration (see Informed Consent).
* Females and males must be willing to use an approved form of birth control while on this study and for 2 weeks after completion.
* Patients of ages 18-80 are eligible provided they have stage IV melanoma and are negative for BRAF or have failed BRAF inhibitor treatment or if they have failed or are intolerant to other established therapy known to provide clinical benefit for their condition or if they have been adequately consented and agreed to forgo FDA approved clinically meaningful therapy.

Exclusion Criteria:

* Failure to meet any of the criteria set forth in Inclusion Criteria.
* Inability to give informed consent because of psychiatric problems, or complicated medical problems.
* Serious concurrent medical problems, uncontrolled infections, or disseminated intravascular coagulopathy (DIC).
* Preexisting cardiovascular disease, the only exception being well controlled essential hypertension with a sitting B.P. of <155 systolic and <90 diastolic without any evidence of structural heart disease or one episode of myocardial infarction > 8 months ago. A past history of the any of the following are exclusions:

  * Congestive heart failure,
  * Atrial fibrillation,
  * Pulmonary hypertension,
  * Anticoagulant drug therapy,
  * Thromboembolic events,
  * Cardiomyopathy or a myocardial infarction within the past 8 months. Referring physicians will be asked to verify that their referred patients do not have these exclusionary histories listed in 3.2 and a copy of this verification must be sent to the Sponsor before the Sponsor will approve of enrollment. Because beta-blockers have been associated with adverse events during anaphylactic reactions and because such reactions can occur with IV infusions of proteins such as the study drug, the sponsor requires that patients receiving beta-blockers for hypertension be converted to another anti-hypertensive reagent 2-3 weeks prior to receiving the study drug. Angiotensin inhibitors, angiotensin receptor blockers and calcium channel blockers are all acceptable.
* Pregnant or nursing women will be excluded from study.
* History of congestive heart failure.
* History of cirrhosis of the liver.
* Prior treatment with alemtuzumab (Campath) or similar agents or procedures that depress blood T cell counts to below 50% of the lower limit of normal.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-02 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Clinical Response primary outcome measure is the change in Progression Free Survival time (PFS). | 2 months, then at least every 3 months post treatment or until disease progression (maximum 36 months)
  The PFS time will be determined as the time from enrollment until the first adverse event (i.e., disease progression or death due to any cause).

SECONDARY OUTCOMES:
Changes in Clinical Response Rates | 2 months, then at least every 3 months post treatment or until disease progression (maximum 36 months)
  Changes in clinical response rates (complete, partial, and sustained) along with 95% estimated confidence intervals compared to the historical record of Pembrolizumab and local palliative radiation. Disease progression and efficacy response will be determined using RECIST 1.1. At a minimum, CT scans of the chest, abdomen, and pelvis will be performed at study entry, at 2 months, and, if a response or stable disease, at least every 3 months (±7 days) for up to 1 year after the last dose of study drug, and/or at any time there is clinical evidence of disease progression, to evaluate disease status (assessed up to 36 months).
Tolerability to Treatment | 2 months, then at least every 3 months post treatment or until disease progression (maximum 36 months)
  Determine the tolerability of A-dmDT390-bisFv(UCHT1) at a total dose of 20 μg/kg when combined with Pembrolizumab and local palliative radiation towards metastatic lesions in stage IV melanoma as a percentage of patients experiencing serious adverse events. The cumulative number of CTCAE grade 3 or 4 toxic events either from lab data or clinical findings will be monitored. Multiple measurements will be aggregated to arrive at one reported value (e.g., Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment).
Overall Survival, OS | 2 months, then at least every 3 months post treatment (maximum 36 months)
  The OS time will be determined as the time from enrollment until death or last follow-up evaluation, assessed up to 36 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Chesney, MD, PhD, Principal Investigator — James Graham Brown Cancer
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schumacher TN, Schreiber RD. Neoantigens in cancer immunotherapy. Science. 2015 Apr 3;348(6230):69-74. doi: 10.1126/science.aaa4971. PMID 25838375
- [Background] Blake SJ, Ching AL, Kenna TJ, Galea R, Large J, Yagita H, Steptoe RJ. Blockade of PD-1/PD-L1 promotes adoptive T-cell immunotherapy in a tolerogenic environment. PLoS One. 2015 Mar 5;10(3):e0119483. doi: 10.1371/journal.pone.0119483. eCollection 2015. PMID 25741704
- [Background] Ahmadzadeh M, Johnson LA, Heemskerk B, Wunderlich JR, Dudley ME, White DE, Rosenberg SA. Tumor antigen-specific CD8 T cells infiltrating the tumor express high levels of PD-1 and are functionally impaired. Blood. 2009 Aug 20;114(8):1537-44. doi: 10.1182/blood-2008-12-195792. Epub 2009 May 7. PMID 19423728
- [Result] Frankel AE, Woo JH, Ahn C, Foss FM, Duvic M, Neville PH, Neville DM. Resimmune, an anti-CD3epsilon recombinant immunotoxin, induces durable remissions in patients with cutaneous T-cell lymphoma. Haematologica. 2015 Jun;100(6):794-800. doi: 10.3324/haematol.2015.123711. Epub 2015 Mar 20. PMID 25795722